CLINICAL TRIAL: NCT00408733
Title: Evaluating a Low-Literacy Discharge Medication Education Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Kristina Cordasco, UCLA
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: G06-09-104-01
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2007-12

CONDITIONS: Congestive Heart Failure; Coronary Artery Disease
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): Intervention
  Interventions: Other: Medication Education Tool

INTERVENTIONS:
Other: Medication Education Tool — Picture and Icon-based Customizable Educational Tool
  Arms: 2

SUMMARY:
Recent studies have demonstrated that patients sub-optimally understand hospital discharge medication instructions Health literacy has been shown to be an important factor in patient understanding of medical information , and following medication instructions.

The primary aim of this project is to test the efficacy of a low-literacy discharge medication education tool on medication adherence, and patient knowledge and understanding of inpatient discharge medications, in a low-income population with low health literacy levels. This evaluation is a prospective trial with patients randomly assigned to either receiving this tool or receiving the current standard of care. Given the complexity of the discharge medication regimen for the conditions of congestive heart failure (CHF) and coronary artery disease (CAD), and the proven effectiveness of these medications in the post discharge period, this trial will focus on the subpopulation of patients hospitalized with these two conditions.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria will be:

* 18 years of age or greater
* Admission to the internal medical or cardiology services at LAC/USC Medical Center
* Discharge directly from the medical service to home
* During admission, being evaluated or treated for congestive heart failure or coronary artery disease.

Patient Exclusion criteria :

* Moderate or severe cognitive dysfunction
* Severe psychiatric disability such that the patient has, or there is an application for, a conservator, or any psychiatric illness with current psychotic features
* Not having speaking proficiency in either English or Spanish language.
* If the patient was previously enrolled in the study on a prior hospitalization, he or she will also be excluded.

Nurse Inclusion Criteria:

* Performing the patient education at hospital discharge for a patient enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Self-Reported Medication Adherence | 2 & 4 weeks post discharge

SECONDARY OUTCOMES:
Medication Knowledge, Patient Satisfaction & Self-Efficacy, Readmissions and Emergency Department Visits | 2weeks -8weeks post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Cordasco, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- Los Angeles County/ USC Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Cordasco KM, Asch SM, Bell DS, Guterman JJ, Gross-Schulman S, Ramer L, Elkayam U, Franco I, Leatherwood CL, Mangione CM. A low-literacy medication education tool for safety-net hospital patients. Am J Prev Med. 2009 Dec;37(6 Suppl 1):S209-16. doi: 10.1016/j.amepre.2009.08.018. PMID 19896021